CLINICAL TRIAL: NCT01496209
Title: REgenerative CardiOsphere iNjection to STRengthen dysfUnCTional Hearts
Acronym: RECONSTRUCT
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Eduardo Marban, MD, PhD, Director, Heart Institute, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RECONSTRUCT
Record Dates: First submitted 2011-12-19; First posted 2011-12-21 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Ischemic Cardiomyopathy; Chronic Ischemic Cardiomyopathy
Keywords: Infarction; Myocardial Infarction; Ventricular Dysfunction, Left; Heart Disease; Cardiovascular Disease; Chronic Ischemia
MeSH Terms: conditions — Infarction; Myocardial Infarction; Ventricular Dysfunction, Left; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo control (Sham Comparator)
  Interventions: Biological: Endomyocardial injections of vehicle only.
- Group: Cardiosphere Treatment (Experimental): Biological: Allogeneic Human Cardiospheres (allogeneic CSps or alloCSps), a 3D micro-tissue heart-derived cell therapy product. Subjects will receive 150 million cell-equivalents of alloCSps via endomyocardial injection (10 million per site at 15 peri-infarct sites)
  Interventions: Biological: Endomyocardial injections of allogeneic Human CSps

INTERVENTIONS:
Biological: Endomyocardial injections of allogeneic Human CSps — NOGA electromechanical mapping and endomyocardial injections at 15 peri-infarct sites, via NOGA MYOSTAR catheter, of Allogeneic Human CSps.
  Other Names: Biological: Allogeneic Human CSps (or alloCSps)
  Arms: Group: Cardiosphere Treatment
Biological: Endomyocardial injections of vehicle only. — NOGA electromechanical mapping and endomyocardial injections at 15 peri-infarct sites, via NOGA MYOSTAR catheter, of placebo.
  Arms: Placebo control

SUMMARY:
A double blinded and placebo-controlled, dose escalation, single-center safety and preliminary efficacy study of cardiospheres delivered via NOGA MYOSTAR injection catheter in subjects with chronic ischemic cardiomyopathy. The objective is to achieve and document myocardial regeneration in patients with chronic scar.

ELIGIBILITY:
Inclusion Criteria:

* Adults with ischemic cardiomyopathy (EF >10 and <40% by functional imaging [ECHO, CT, MRI, contrast ventriculography])
* Symptomatic heart failure of NYHA Class 2 or 3
* History of prior remote (>3 mo) myocardial infarction and/or documented obstructive coronary artery disease with corresponding dysfunctional segments by functional imaging
* Age > 18 years
* Ability to provide informed consent and follow-up with protocol procedures

Exclusion Criteria:

* Documented myocardial infarction within 3 months (120 days)
* Known or suspected left ventricular thrombus
* Non-cardiovascular disease with life expectancy of < 3 years
* Absence of significant gadolinium-enhanced scar (>10% of LV mass) at baseline MRIc
* Positive panel-reactive antibodies (PRA)
* Need for further revascularization clinically indicated at the time the patient is assessed for participation in the clinical trial. This will be determined by a cardiologist who is not an investigator in the clinical trial. No further revascularization may be indicated by no arteries with significant stenosis, the location, and extent of any stenosis may not be suitable for angioplasty, the distal vessels may not be suitable for placement of bypass grafts, and/or the patient declines angioplasty or bypass surgery.
* NYHA IV heart failure
* History of aortic stenosis/insufficiency
* Requirement for chronic immunosuppressive therapy
* Participation in an on-going protocol studying an experimental drug or device
* Diagnosis of congenital or genetically-transmitted cardiomyopathy
* Current alcohol or drug abuse because of anticipated difficulty in complying with protocol-related procedures
* Pregnancy or child-bearing potential without use of effective contraception. Men intending to "father" children are also excluded.
* Human Immunodeficiency virus infection
* Viral hepatitis
* Uncontrolled diabetes and/or hemoglobin A1C > 8.5%
* Abnormal liver function (SGPT > 3 times the upper reference range) and/or hematology (hematocrit <25%, WBC <3000, Platelets <100,000) studies without a reversible, identifiable cause
* Ventricular tachycardia or fibrillation not associated with an acute ischemic episode
* Canadian Cardiovascular Society Angina Class 3 or 4
* History of cardiac tumor or cardiac tumor demonstrated or suspected on MRI other imaging modality
* Previous stem cell therapy/treatment
* Individuals who are not fluent in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Marban, MD, PhD, Principal Investigator — Cedars-Sinai Medical Center, Heart Institute
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States